CLINICAL TRIAL: NCT00285129
Title: Primary Ceramic-on-Ceramic Total Hip Replacement Versus Metal-on-Metal Hip Resurfacing in Young Active Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004/338
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Indications for a Total Hip Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ceramic-on-ceramic total hip replacement versus metal-on-metal hip resurfacing

SUMMARY:
Comparison of the functional result and speed of rehabilitation between two types of hip prostheses: primary ceramic-on-ceramic total hip replacement versus metal-on-metal hip resurfacing.

ELIGIBILITY:
Inclusion Criteria:

* Total hip replacement

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2004-01; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Functional result
Speed of rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Rene Verdonk, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be